CLINICAL TRIAL: NCT02317016
Title: A Phase I, Open-Label, Non-Randomised, Multicentre Study to Assess the Effect of AZD9291 on the Pharmacokinetics of Rosuvastatin (a Sensitive BCRP Substrate) in Patients With EGFRm Positive NSCLC Whose Disease Has Progressed on an EGFR TKI
Brief Title: Study to Assess the Effect of AZD9291 on the Blood Levels of Rosuvastatin, in Patients With EGFRm+ Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5160C00019
Record Dates: First submitted 2014-12-11; First posted 2014-12-15 (Estimated); Results first posted 2016-07-14 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2018-06

CONDITIONS: Non Small Cell Lung Cancer
Keywords: oncology; cancer; non small cell lung cancer; anticancer drug; pharmacokinetics; AZD9291; rosuvastatin; EGFR genes
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AZD9291 and rosuvastatin (Experimental): Sequential treatments of rosuvastatin alone followed by AZD9291 alone, followed by rosuvastatin + AZD9291.
  Interventions: Procedure: Pharmacokinetic sampling - AZD9291; Drug: AZD9291 tablet dosing; Drug: Rosuvastatin; Procedure: Pharmacokinetic sampling - rosuvastatin; Procedure: Pharmacokinetic sampling - AZ5140 and AZ7550

INTERVENTIONS:
Procedure: Pharmacokinetic sampling - AZD9291 — Blood sampling to measure AZD9291
Drug: AZD9291 tablet dosing — Part A: AZD9291 80mg tablet taken from Days 4 to 35. Part B: AZD9291 80mg tablet taken daily for 12 months.
Drug: Rosuvastatin — Rosuvastatin (BCRP substrate) 20mg taken once daily on Days 1 and 32 (Part A) .
Procedure: Pharmacokinetic sampling - rosuvastatin — Blood sampling to measure rosuvastatin levels
Procedure: Pharmacokinetic sampling - AZ5140 and AZ7550 — Blood samples to measure levels of AZ5140 and AZ7550

SUMMARY:
This is a Phase I, open-label, 2-part study in patients with a confirmed diagnosis of epidermal growth factor receptor (EGFR) mutation positive (EGFRm+) non-small cell lung cancer (NSCLC), who have progressed following prior therapy with an approved EGFR tyrosine kinase inhibitor (TKI) agent.

Part A will assess the effect of AZD9291 on the pharmacokinetic (PK) parameters of rosuvastatin, following multiple oral dosing of AZD9291 in the fasted state.

Part B will allow patients further access to AZD9291 after the PK phase (Part A) and will provide for additional safety data collection. All patients from Part A who completed treatment may continue to receive AZD9291 80 mg once daily as a single agent until: disease progression; they are no longer deriving clinical benefit; or any other reason.

ELIGIBILITY:
For inclusion in the study patients must fulfil the following criteria:

1. Male or female, aged at least 18 years.
2. Histological or cytological confirmation diagnosis of NSCLC.
3. Radiological documentation of disease progression while on a previous continuous treatment with an EGFR TKI, eg, gefitinib, erlotinib or afatinib. In addition, other lines of therapy may have been given. All patients must have documented radiological progression on the last treatment administered prior to enrolling in the study.
4. Confirmation that the tumour harbours an EGFR mutation known to be associated with EGFR TKI sensitivity (including G719X, exon 19 deletion, L858R, L861Q).
5. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1 with no deterioration over the previous 2 weeks (Appendix G).
6. Patients must have a life expectancy of ≥12 weeks as estimated at the time of screening.
7. Females should be using adequate contraceptive measures and must have a negative pregnancy test prior to start of dosing if of child-bearing potential, or must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening: Post-menopausal defined as aged more than 50 years and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatments; Women under 50 years old would be considered post-menopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments and with luteinising hormone (LH) and follicle stimulating hormone (FSH) levels in the post-menopausal range for the institution; Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy, but not tubal ligation.
8. Patients are willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.
9. Male patients should be willing to use barrier contraception, ie, condoms.

Exlusion Criteria:

1. Participation in another clinical study with an IP in last 14 days (or longer depending on the defined characteristics of the agents used).
2. Any patient of Asian ethnicity or has a parent who is of Asian ethnicity (eg, Chinese, Filipino, Japanese, Korean and Vietnamese). If only a grandparent is Asian, this is acceptable. Asian Indians are acceptable.
3. Treatment w/ any of the following: an EGFR TKI (eg, erlotinib, gefitinib or afatinib) within 8 days or approx. 5 x half-life, whichever is the longer, of the first dose of study treatment; Any cytotoxic chemotherapy, investigational agents or other anticancer drugs from a previous treatment regimen or clinical study within 14 days of the first dose of study treatment; Major surgery (excluding placement of vascular access) w/in 4 weeks of the 1st dose of study treatment; Radiotherapy with a limited field of radiation for palliation w/in 1 week of the first dose of study treatment, with the exception of patients receiving radiation to more than 30% of bone marrow or with a wide field of radiation which must be completed w/in 4 weeks of the 1st dose of study treatment; Patients currently receiving (or unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be potent inhibitors of CYP3A4 (at least 1 week prior) and potent inducers of CYP3A4 (at least 3 week prior). All patients must avoid concomitant use of any medications, herbal supplements and/or ingestion of foods with known inducer/inhibitory effects on CYP3A4.
4. Unresolved toxicities from prior therapy > CTCAE Grade 1 at the study start besides alopecia and Grade 2, prior platinum-therapy related neuropathy.
5. Any intake of grapefruit, grapefruit juice, Seville oranges, Seville orange marmalade, or other products containing grapefruit or Seville oranges within 7 days of the first administration of the IP until the final PK sample collection on Day 35 of Part A.
6. Spinal cord compression or brain metastases unless asymptomatic, stable and not requiring steroids for at least 4 weeks prior to start of study treatment.
7. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the PI's opinion makes it undesirable for the patient to participate in the study or which would jeopardise compliance with the protocol, or active infection including hep B, hep C and HIV. Screening for chronic conditions is not required.
8. Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values: ANC<1.5 x 10^9/L; Platelet count <100 x 10^9/L; Haemoglobin <90 g/L; ALT >2.5 times ULN if no demonstrable liver metastases or >5 times ULN in the presence of liver metastases; AST >2.5 times ULN if no demonstrable liver metastases or >5 times ULN in the presence of liver metastases; Total bilirubin >1.5 times ULN if no liver metastases or >3 times ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinaemia) or liver metastases; Creatinine >1.5 times ULN concurrent with creatinine clearance <50 mL/min (measured or calculated by Cockcroft and Gault equation); confirmation of creatinine clearance is only required when creatinine is >1.5 times ULN.
9. Any of the following cardiac criteria: Mean resting corrected QT interval corrected for heart rate using Fridericia's correction factor (QTcF) >470 msec obtained from 3 ECGs; Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG eg, complete left bundle branch block, third degree heart block, second degree heart block, PR interval >250 msec; Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age or any concomitant medication known to prolong the QT interval
10. Patients unable to swallow orally administered medication or patients with gastrointestinal disorders or significant gastrointestinal resection likely to interfere with the absorption of AZD9291.
11. Past medical history of ILD, drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD.
12. Women who are breastfeeding.
13. Patients with a known hypersensitivity to AZD9291 or rosuvastatin or any of the excipients of the products.
14. Concomitant medication contraindicated for use with rosuvastatin due to drug interaction and/or associated with increased risk of rhabdomyolysis (including, but not limited to): fibrates (eg, gemfibrozil, fenofibrate), niacin, cyclosporine, lopinavir/ritonavir or atazanavir/ritonavir and colchinine.
15. Past medical history of drug-related rhabdomyolysis and/or myalgia.
16. Use of 3-hydroxy-3-methyl-glutaryl coenzyme A-reductase inhibitors, such as lovastatin and simvastatin (Part A only).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-03-10 (Actual); Primary Completion 2015-07-11 (Actual); Study Completion 2018-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Serban Ghiorghiu, MSD, Study Director — AstraZeneca
Locations (10):
- Research Site, Fairfax, Virginia, United States
- France (3):
  - Research Site, Bordeaux
  - Research Site, Montpellier
  - Research Site, Rennes
- Spain (4):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Seville
- United Kingdom (2):
  - Research Site, London
  - Research Site, Manchester

REFERENCES:
- [Derived] Harvey RD, Aransay NR, Isambert N, Lee JS, Arkenau T, Vansteenkiste J, Dickinson PA, Bui K, Weilert D, So K, Thomas K, Vishwanathan K. Effect of multiple-dose osimertinib on the pharmacokinetics of simvastatin and rosuvastatin. Br J Clin Pharmacol. 2018 Dec;84(12):2877-2888. doi: 10.1111/bcp.13753. Epub 2018 Oct 10. PMID 30171779

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled: 10 March 2015; Last Subject Last Visit Part A: 11 July 2015 and Part B: 11 July 2016. Study performed at 14 sites across North America and Western Europe. Part A assessed effect of AZD9291 on PK of rosuvastatin following multiple oral dosing; Part B allowed subjects further access to AZD9291 and additional safety data.
Groups:
- Rosuvastatin and AZD9291 (Part A); AZD9291 Alone (Part B): In Part A of the study, sequential treatments of rosuvastatin alone, followed by AZD9291 alone, followed by rosuvastatin + AZD9291. Each patient received 20 mg single oral doses of rosuvastatin on Day 1 and Day 32, and 80 mg oral doses of AZD9291 tablets once daily for 31 days (Days 4 to 34).
  In Part B of the study, each patient received 80 mg oral AZD9291 tablet formulation once daily, for the duration of their participation.
Period: Part A: Day 1-3 (Rosuvastatin Alone)
Arm/Group | Rosuvastatin and AZD9291 (Part A); AZD9291 Alone (Part B)
Started | 44
Completed | 44
Not Completed | 0
Period: Part A: Day 4-31 (AZD9291 Alone)
Arm/Group | Rosuvastatin and AZD9291 (Part A); AZD9291 Alone (Part B)
Started | 44
Completed | 43
Not Completed | 1
Not completed — Adverse Event | 1
Period: Part A: Day 32-34 (Rosuvastatin+AZD9291)
Arm/Group | Rosuvastatin and AZD9291 (Part A); AZD9291 Alone (Part B)
Started | 43
Completed | 41
Not Completed | 2
Not completed — Condition under investigation worsened | 1
Not completed — Death | 1
Period: Part B: Day 35 to End Part B (AZD9291)
Arm/Group | Rosuvastatin and AZD9291 (Part A); AZD9291 Alone (Part B)
Started | 42 (41 completed Part A + 1 entered Part B without completing Part A (due to AE) = 42 started Part B)
Completed | 11
Not Completed | 31
Not completed — Condition under investigation worsened | 23
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 2
Not completed — Death | 5

BASELINE CHARACTERISTICS:
Population: All patients in the safety analysis set who received at least one dose of AZD9291 or rosuvastatin (n = 44) were included in the baseline analysis.
Arm/Group | Rosuvastatin and AZD9291 (Part A); AZD9291 Alone (Part B)
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (11.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 41
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Maximum Plasma Concentration (Cmax) for Rosuvastatin After a Single Dose Alone and in Combination With AZD9291
Description: Rate and extent of absorption of rosuvastatin by assessment of Cmax. Single rosuvastatin doses were first without, then with AZD9291 (Day 1 [Period 1] and Day 32 [Period 3], respectively).
Time Frame: Blood samples collected on Days 1 and 32 at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 60, and 72 hours post rosuvastatin dose in Part A.
Population: The PK analysis set included all dosed patients who had at least 1 quantifiable plasma concentration collected post-dose without any important deviations or events that would exclude the patient.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per millilitre (ng/mL)
Groups:
- Rosuvastatin Alone (Period 1 [Day 1]): Rosuvastatin 20 mg single oral dose on Day 1 (Part A). Rosuvastatin was administered fasted from at least 2 hours before dosing to at least 2 hours after dosing. Water was allowed as desired except for 1 hour before and after dose.
- AZD9291 + Rosuvastatin (Period 3 [Day 32]): Steady state AZD9291 80 mg in combination with rosuvastatin 20 mg single oral dose on Day 32 (Part A). The Day 32 treatment (AZD9291 plus rosuvastatin) could occur within a window of ±2 days. Treatment was administered fasted from at least 2 hours before dosing to at least 2 hours after dosing. Water was allowed as desired except for 1 hour before and after dose. Previously, patients had received AZD9291 80 mg once daily for 28 days during Period 2 (Days 4 to 31), and after Day 32 in Period 3 (Days 33 and 34) patients also received AZD9291 80 mg once daily doses.
Arm/Group | Rosuvastatin Alone (Period 1 [Day 1]) | AZD9291 + Rosuvastatin (Period 3 [Day 32])
Number analyzed (Participants) | 42 | 39
nanogram per millilitre (ng/mL) | 13.96 (66.7) | 24.03 (70.5)
Statistical Analysis 1: Comparison: Rosuvastatin Alone (Period 1 [Day 1]) vs AZD9291 + Rosuvastatin (Period 3 [Day 32]); Natural log-transformed Cmax values were compared between treatments using a mixed effects analysis of variance (ANOVA) with treatment as a fixed effect and patient as a random effect. It was assumed the within-patient coefficient of variation for rosuvastatin in both area under the plasma concentration-time curve (AUC) and Cmax was 41%. No change in the exposure for rosuvastatin when given with AZD9291 was also assumed; Test type: Non-Inferiority or Equivalence — No effect on the PK of rosuvastatin after co-administration of AZD9291 was concluded if the 2-sided 90% confidence intervals (CIs) for the ratios of rosuvastatin AUC and Cmax were within the range of 70% to 143%; Geometric least-squares (LS) mean ratio = 171.92, 90% CI 2-sided [145.94 to 202.53] — AZD9291+ rosuvastatin / rosuvastatin alone (Day 32 versus Day 1)

2. Primary Outcome: Assessment of AUC From Time Zero Extrapolated to Infinity for Rosuvastatin After a Single Dose Alone and in Combination With AZD9291
Description: Rate and extent of absorption of rosuvastatin by assessment of AUC from time zero extrapolated to infinity. Single rosuvastatin doses were first without, then with AZD9291 (Day 1; Period 1 and Day 32; Period 3, respectively).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng * h o u r per mL (ng*h/mL )
Arm/Group | Rosuvastatin Alone (Period 1 [Day 1]) | AZD9291 + Rosuvastatin (Period 3 [Day 32])
Number analyzed (Participants) | 31 | 32
ng * h o u r per mL (ng*h/mL ) | 139.1 (49.0) | 185.7 (60.9)
Statistical Analysis 1: Comparison: Rosuvastatin Alone (Period 1 [Day 1]) vs AZD9291 + Rosuvastatin (Period 3 [Day 32]); Natural log-transformed AUC values were compared between treatments using a mixed effects ANOVA with treatment as a fixed effect and patient as a random effect. It was assumed the within-patient coefficient of variation for rosuvastatin in both AUC and Cmax was 41%. No change in the exposure for rosuvastatin when given with AZD9291 was also assumed; Test type: Non-Inferiority or Equivalence — No effect on the PK of rosuvastatin after co-administration of AZD9291 was concluded if the 2-sided 90% CIs for the ratios of rosuvastatin AUC and Cmax were within the range of 70% to 143%; Geometric LS Mean Ratio = 134.63, 90% CI 2-sided [115.41 to 157.07] — AZD9291+ rosuvastatin / rosuvastatin alone (Day 32 versus Day 1)

3. Secondary Outcome: Assessment of Time to Maximum Plasma Concentration (Tmax) for Rosuvastatin After a Single Dose Alone and in Combination With AZD9291
Description: Rate and extent of absorption of rosuvastatin by assessment of tmax. Single rosuvastatin doses were first without, then with AZD9291 (Day 1; Period 1 and Day 32; Period 3, respectively).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | Rosuvastatin Alone (Period 1 [Day 1]) | AZD9291 + Rosuvastatin (Period 3 [Day 32])
Number analyzed (Participants) | 42 | 39
h | 2.05 [0.48 to 5.95] | 2.07 [0.47 to 6.00]

4. Secondary Outcome: Assessment of Area Under the Plasma Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration at Time "t" (AUC0-t) for Rosuvastatin After a Single Dose Alone and in Combination With AZD9291
Description: Rate and extent of absorption of rosuvastatin by assessment of AUC0-t. Single rosuvastatin doses were first without, then with AZD9291 (Day 1; Period 1 and Day 32; Period 3, respectively).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Rosuvastatin Alone (Period 1 [Day 1]) | AZD9291 + Rosuvastatin (Period 3 [Day 32])
Number analyzed (Participants) | 42 | 37
ng*h/mL | 130.6 (51.1) | 183.7 (58.3)

5. Secondary Outcome: Assessment of Apparent Plasma Clearance (CL/F) for Rosuvastatin After a Single Dose Alone and in Combination With AZD9291
Description: Rate and extent of absorption of rosuvastatin by assessment of CL/F. Single rosuvastatin doses were first without, then with AZD9291 (Day 1; Period 1 and Day 32; Period 3, respectively).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litre / h (L/h)
Arm/Group | Rosuvastatin Alone (Period 1 [Day 1]) | AZD9291 + Rosuvastatin (Period 3 [Day 32])
Number analyzed (Participants) | 31 | 32
Litre / h (L/h) | 143.8 (49.0) | 107.7 (60.9)

6. Secondary Outcome: Assessment of Apparent Volume of Distribution (Vz/F) for Rosuvastatin After a Single Dose Alone and in Combination With AZD9291
Description: Rate and extent of absorption of rosuvastatin by assessment of Vz/F. Single rosuvastatin doses were first without, then with AZD9291 (Day 1; Period 1 and Day 32; Period 3, respectively).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Rosuvastatin Alone (Period 1 [Day 1]) | AZD9291 + Rosuvastatin (Period 3 [Day 32])
Number analyzed (Participants) | 31 | 32
L | 3890 (65.0) | 2874 (77.9)

7. Secondary Outcome: Assessment of Terminal Elimination Half-life (t1/2[lambda_z]) for Rosuvastatin After a Single Dose Alone and in Combination With AZD9291
Description: Rate and extent of absorption of rosuvastatin by assessment of t1/2(lambda_z). Single rosuvastatin doses were first without, then with AZD9291 (Day 1; Period 1 and Day 32; Period 3, respectively).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Rosuvastatin Alone (Period 1 [Day 1]) | AZD9291 + Rosuvastatin (Period 3 [Day 32])
Number analyzed (Participants) | 31 | 32
h | 18.75 (29.5) | 18.51 (37.4)

8. Secondary Outcome: Assessment of Area Under the Plasma Concentration-time Curve During the Dosing Interval (AUCtau) for AZD9291, and AZ5104 and AZ7550 (Metabolites) Following Administration of AZD9291 and Rosuvastatin Together
Description: Rate and extent of absorption for AZD9291, and AZ5104 and AZ7550 (metabolites) by assessment of AUCtau. AZD9291 doses were first without, then with rosuvastatin (Days 4 to 31; Period 2 and Day 32; Period 3, respectively).
Time Frame: Blood samples collected pre-dose on Days 11, 18, and 25 and on Day 32 at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, and 24 hours post AZD9291 dose in Part A.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomolar * h (nM*h)
Arm/Group | AZD9291 + Rosuvastatin (Period 3 [Day 32])
Number analyzed (Participants) | 37
nanomolar * h (nM*h)
  AZD9291 AUCtau | 15800 (45.0)
  AZ5104 AUCtau | 1655 (62.1)
  AZ7550 AUCtau | 1418 (44.7)

9. Secondary Outcome: Assessment of Maximum Plasma Concentration at Steady State (Css,Max) for AZD9291, and AZ5104 and AZ7550 (Metabolites) Following Administration of AZD9291 and Rosuvastatin Together
Description: Rate and extent of absorption for AZD9291, and AZ5104 and AZ7550 (metabolites) by assessment of Css,max after multiple dosing. AZD9291 doses were first without, then with rosuvastatin (Days 4 to 31; Period 2 and Day 32; Period 3, respectively).
Time Frame: as for outcome 8
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | AZD9291 + Rosuvastatin (Period 3 [Day 32])
Number analyzed (Participants) | 37
nM
  AZD9291 Css,max | 897.9 (47.2)
  AZ5104 Css,max | 86.20 (60.3)
  AZ7550 Css,max | 73.73 (47.3)

10. Secondary Outcome: Assessment of Time to Reach Maximum Plasma Concentration at Steady State (Tss,Max) for AZD9291, and AZ5104 and AZ7550 (Metabolites) Following Administration of AZD9291 and Rosuvastatin Together
Description: Rate and extent of absorption for AZD9291, and AZ5104 and AZ7550 (metabolites) by assessment of tss,max after multiple dosing. AZD9291 doses were first without, then with rosuvastatin (Days 4 to 31; Period 2 and Day 32; Period 3, respectively).
Time Frame: as for outcome 8
Population: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | AZD9291 + Rosuvastatin (Period 3 [Day 32])
Number analyzed (Participants) | 37
h
  AZD9291 tss,max | 5.00 [2.00 to 8.17]
  AZ5104 tss,max | 5.00 [0.50 to 24.33]
  AZ7550 tss,max | 5.05 [1.50 to 12.05]

11. Secondary Outcome: Assessment of Minimum Plasma Concentration at Steady State (Css,Min) for AZD9291, and AZ5104 and AZ7550 (Metabolites) Following Administration of AZD9291 and Rosuvastatin Together
Description: Rate and extent of absorption for AZD9291, and AZ5104 and AZ7550 (metabolites) by assessment of Css,min over the dosing interval. AZD9291 doses were first without, then with rosuvastatin (Days 4 to 31; Period 2 and Day 32; Period 3, respectively).
Time Frame: as for outcome 8
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | AZD9291 + Rosuvastatin (Period 3 [Day 32])
Number analyzed (Participants) | 37
nM
  AZD9291 Css,min | 485.6 (47.3)
  AZ5104 Css, min | 54.60 (63.6)
  AZ7550 Css, min | 46.46 (46.3)

12. Secondary Outcome: Assessment of Apparent Plasma Clearance at Steady State (CLss/F) for AZD9291 Following Administration of AZD9291 and Rosuvastatin Together
Description: Rate and extent of absorption for AZD9291 by assessment of CLss/F after multiple dosing. AZD9291 doses were first without, then with rosuvastatin (Days 4 to 31; Period 2 and Day 32; Period 3, respectively).
Time Frame: as for outcome 8
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | AZD9291 + Rosuvastatin (Period 3 [Day 32])
Number analyzed (Participants) | 37
L/h | 10.14 (45.0)

13. Secondary Outcome: Assessment of the Metabolite to Parent Ratios of Css,Max (MRCss,Max) for AZ5104 and AZ7550 Following Administration of AZD9291 and Rosuvastatin Together
Description: Assessment of MRCss,max for AZ5104 and AZ7550 (calculated as AZ5104 to AZD9291 and AZ7550 to AZD9291) after multiple dosing. AZD9291 doses were first without, then with rosuvastatin (Days 4 to 31; Period 2 and Day 32; Period 3, respectively).
Time Frame: as for outcome 8
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | AZD9291 + Rosuvastatin (Period 3 [Day 32])
Number analyzed (Participants) | 37
Ratio
  AZ5104 Css,max / AZD9291 Css,max | 0.09599 (28.2)
  AZ7550 Css,max / AZD9291 Css,max | 0.08212 (31.7)

14. Secondary Outcome: Assessment of the Metabolite to Parent Ratios of AUCtau (MRAUCtau) for AZ5104 and AZ7550 Following Administration of AZD9291 and Rosuvastatin Together
Description: Assessment of MRAUCtau for AZ5104 and AZ7550 (calculated as AZ5104 to AZD9291 and AZ7550 to AZD9291) after multiple dosing. AZD9291 doses were first without, then with rosuvastatin (Days 4 to 31; Period 2 and Day 32; Period 3, respectively).
Time Frame: as for outcome 8
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | AZD9291 + Rosuvastatin (Period 3 [Day 32])
Number analyzed (Participants) | 37
Ratio
  AZ5104 AUCtau / AZD9291 AUCtau | 0.1048 (28.1)
  AZ7550 AUCtau / AZD9291 AUCtau | 0.08971 (33.6)

ADVERSE EVENTS:
Time Frame: Approximately 1 month for Part A; up to approximately 14 months for Part B and approximately 15 months for Overall (Parts A and B combined).
Description: Part A: Adverse events (AEs) collected from day of first dose until day prior to first dose in Part B (Day 35), or until 30 days after last dose if discontinued in Part A.
  Part B: AEs collected from day of first dose in Part B until 30 days after last dose, or until last dose in Part B for those entering continued access phase (CAP).
Groups:
- Overall Safety Population: Parts A and B of the study combined.
- Part A Safety Population: In Part A of the study, each patient received 80 mg oral doses of AZD9291 tablets once daily for 31 days (Days 4 to 34) and single 20 mg oral doses of rosuvastatin on Day 1 and Day 32.
- Part B Safety Population: In Part B of the study, each patient received 80 mg oral AZD9291 tablet formulation once daily, for the duration of their participation.
Arm/Group | Overall Safety Population | Part A Safety Population | Part B Safety Population
Serious Adverse Events (participants affected / at risk) | 7/44 | 2/44 | 6/42
Other Adverse Events (participants affected / at risk) | 40/44 | 34/44 | 29/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Safety Population (N=44) | Part A Safety Population (N=44) | Part B Safety Population (N=42)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pneumonia pseudomonal (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Safety Population (N=44) | Part A Safety Population (N=44) | Part B Safety Population (N=42)
Anaemia (Blood and lymphatic system disorders) | 4 (6) | 3 (3) | 2 (3)
Constipation (Gastrointestinal disorders) | 6 (7) | 4 (4) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 13 (27) | 9 (12) | 9 (15)
Vomiting (Gastrointestinal disorders) | 3 (5) | 2 (2) | 2 (3)
Fatigue (General disorders) | 8 (9) | 5 (5) | 3 (4)
Blood creatine phosphokinase increased (Investigations) | 3 (3) | 0 (0) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (9) | 2 (2) | 5 (7)
Vertigo (Ear and labyrinth disorders) | 3 (5) | 2 (2) | 3 (3)
Dry eye (Eye disorders) | 3 (3) | 0 (0) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 7 (8) | 4 (4) | 3 (4)
Stomatitis (Gastrointestinal disorders) | 3 (4) | 1 (1) | 3 (3)
Asthenia (General disorders) | 9 (12) | 4 (4) | 7 (8)
Pyrexia (General disorders) | 6 (7) | 3 (3) | 4 (4)
Xerosis (General disorders) | 3 (3) | 1 (1) | 2 (2)
Paronychia (Infections and infestations) | 6 (11) | 1 (1) | 5 (10)
Rhinitis (Infections and infestations) | 4 (4) | 2 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 4 (4) | 3 (3) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 16 (19) | 9 (9) | 9 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 4 (4) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0) | 5 (5)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (4) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (4) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 6 (8) | 2 (2) | 4 (6)
Insomnia (Psychiatric disorders) | 4 (5) | 2 (2) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (15) | 4 (4) | 8 (11)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 8 (8) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1) | 2 (3)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 5 (6) | 2 (2) | 4 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (8) | 1 (1) | 5 (7)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 1 (1)

LIMITATIONS AND CAVEATS:
At end of Part B, the CAP allowed patients to continue receiving AZD9291 if still deriving clinical benefit. No clinical data was databased during the CAP; thus AE data is presented to end of Part B only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator (PI) agrees to collaborate on the contents and formation of any publication and to pay due consideration to comments and opinions offered. AstraZeneca have 30 days for final manuscript review and may require that submission for publication be delayed in order to file patent application.